CLINICAL TRIAL: NCT06991855
Title: Explore the Effects of Nutritional Supplementation of Leucine and Polyunsaturated Fatty Acids on Muscle Health in the Elderly
Brief Title: Effects of Nutritional Supplementation of Leucine and Polyunsaturated Fatty Acids on Muscle Health in the Elderly
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Chang Gung University (Other)
Responsible Party: Principal Investigator, JI-TSENG FANG, Professor, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202500394A3
Record Dates: First submitted 2025-05-27; First posted 2025-05-28 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Sarcopenia; Sarcopenia in Elderly
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Animal-Based Oil Group (Experimental): Participants in this group will supplement with animal-based poly-unsaturated oil. The supplementation will be maintained for 12 weeks.
  Interventions: Dietary Supplement: Animal-Based Oil Group
- Plant-Based Oil Group (Experimental): Participants in this group will supplement with plant-based poly-unsaturated oil. The supplementation will be maintained for 12 weeks.
  Interventions: Dietary Supplement: Plant-Based Oil Group

INTERVENTIONS:
Dietary Supplement: Animal-Based Oil Group — Participants in animal-based oil group will follow a diet in which the primary fat source is animal-based oil. The diet will supplement for 12 weeks.
  Arms: Animal-Based Oil Group
Dietary Supplement: Plant-Based Oil Group — Participants in plant-based oil group will follow a diet in which the primary fat source is plant-based oil. The diet will supplement for 12 weeks.
  Arms: Plant-Based Oil Group

SUMMARY:
Population aging has become a significant global concern, and Taiwan is set to officially enter the "super-aged society" in 2025. As individuals age, various physiological functions gradually decline, including a reduction in muscle mass, which is a key aspect of the aging process.

This interventional study aims to investigate the effects of leucine-rich protein combined with polyunsaturated fatty acid supplementation on middle-aged and elderly individuals (aged 50 and above) who are at high risk for sarcopenia.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 years
* ASMI < 7 kg/m2 in men
* ASMI < 5.7 kg/m2 in women
* Grip strength < 28 kg in men
* Grip strength < 18 kg in women
* Walk speed < 1 m/s

Exclusion Criteria:

* People who are allergic to supplements
* cancer
* heart failure
* kidney disease
* autoimmune disease
* neurodegenerative disease

Ages: 50 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-04-10 (Estimated); Study Completion 2026-04-17 (Estimated)

PRIMARY OUTCOMES:
muscle mass | baseline, 12 weeks
  Utilize Bioelectrical Impedance Analysis (BIA) to measure the Appendicular Skeletal Muscle Mass Index Level (ASMI) (kg/m^2)
muscle function | baseline, 12 weeks
  utilize handgrip dynamometer to measure the hand grip strength (kg).
physical function | baseline, 12 weeks
  To assess the participant's walking speed over a 4-meter distance.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Linkou District, Taiwan

IPD SHARING:
Plan to Share IPD: No